CLINICAL TRIAL: NCT00855660
Title: Investigation of the Effect of Riociguat, Administered as 2.5 mg IR-tablets TID Over 14 Days, on Bone Metabolism in a Randomized, Placebo-controlled, Double-blind, 2-fold Cross-over Design in Healthy Male Subjects
Brief Title: Effect of Riociguat on Bone Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13790; 2008-005569-70 (EudraCT Number)
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Pharmacology, Clinical
Keywords: Bone Metabolism
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riociguat (Active Comparator): Subjects received multiple doses of riociguat (thrice a day) with concomitant administration of ranitidine (once daily) for 14 days
  Interventions: Drug: Riociguat (Adempas, BAY63-2521) immediate release tablet of 2.5 mg
- Placebo (Placebo Comparator): Subjects received placebo (thrice a day) with concomitant administration of ranitidine (once daily) for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) immediate release tablet of 2.5 mg — Riociguat administered in a dose of 2.5 mg (single tablet), thrice daily, over 14 days.
  Arms: Riociguat
Drug: Placebo — Placebo administered as a single tablet, thrice daily, over 14 days.
  Arms: Placebo

SUMMARY:
Investigation of the effect of Riociguat, administered as 2.5 mg IR-tablets TID over 14 days, on bone metabolism.

DETAILED DESCRIPTION:
Clinical pharmacology

ELIGIBILITY:
Inclusion Criteria:

* Healthy male white subjects
* 18 to 45 years of age
* BMI between 18 and 28 kg/m2
* Subjects who are able to understand and follow instructions and who are able to participate in the study for the entire period

Exclusion Criteria:

* Relevant deviation from the normal range in the clinical examination; in clinical chemistry, hematology, or urinalysis
* Resting heart rate in the awake subject below 45 BPM or above 90 BPM
* Systolic blood pressure below 100 mmHg or above 145 mmHg
* Diastolic blood pressure above 95 mmHg
* Relevant pathological changes in the ECG such as a second or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QT / QTc-interval over 450 msec for males
* History of genetic muscle or bone disease of any kind
* Completely sedentary or extremely fit subjects
* Fractures in the preceding 12 months
* Psychiatric diseases
* History of peptic ulcers or relevant gastro-esophageal reflux disease
* Subjects with hypersensitivity to the investigational drug riociguat or ranitidine, or to inactive constituents
* Regular daily consumption of more than half a liter of usual beer or the equivalent quantity of approximately 20 g of alcohol in another form, more than 1 L of xanthine-containing beverages, recent smoking history
* Use of medication within the 2 weeks preceding the study which could have interfered with the investigational drug riociguat or ranitidine
* Subjects with a medical disorder, condition or history of such that would have impaired the subject's ability to participate or complete this study in the opinion of the investigator or the sponsor

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Urinary excretion (over 24 hours) of C-terminal cross-linking telopeptides of type I collagen (CTX) | From Day -01 to 16
  Marker of bone resorption
AUC(0-7) | Pre-dose and up to 7 hours post-dose on Day 0
  Area under the plasma concentration vs time curve (AUC) from zero to 7 hours after single (first) dose for riociguat and its metabolite M-1 (BAY60-4552)
AUC(0-7)ss | Pre-dose and up to 7 hours post-dose on Day 13
  AUC(0-7) at steady state
Cmax | Pre-dose and up to 7 hours post-dose on Day 0
  Maximum drug concentration in plasma after single dose administration for riociguat and its metabolite M-1 (BAY60-4552)
Cmax,ss | Pre-dose and up to 7 hours post-dose on Day 13
  Maximum drug concentration in plasma at steady state during a dosage interval for riociguat and its metabolite M-1 (BAY60-4552)

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 12 weeks
Ctrough | On Days 03 and 08
  Drug concentration in plasma at expected time of minimum (trough) concentration for riociguat and its metabolite M-1 (BAY60-4552)
AUC(0-7)norm | Pre-dose and up to 7 hours post-dose on Day 0
  AUC(0-7) divided by dose per kg body weight for riociguat and its metabolite M-1 (BAY60-4552)
AUC(0-7)ss,norm | Pre-dose and up to 7 hours post-dose on Day 13
  AUC(0-7)ss divided by dose per kg body weight for riociguat and its metabolite M-1 (BAY60-4552)
Cmax,norm | Pre-dose and up to 7 hours post-dose on Day 0
  Maximum drug concentration in plasma after (first) single dose administration divided by dose (mg) per kg body weight for riociguat and its metabolite M-1 (BAY60-4552)
Cmax,ss,norm | Pre-dose and up to 7 hours post-dose on Day 13
  Maximum drug concentration in plasma at steady state during a dosage interval divided by dose (mg) per kg body weight for riociguat and its metabolite M-1 (BAY60-4552)
tmax | Pre-dose and up to 7 hours post-dose on Day 0
  Time to reach maximum drug concentration in plasma after single (first) dose for riociguat and its metabolite M-1 (BAY60-4552)
tmax,ss | Pre-dose and up to 7 hours post-dose on Day 13
  tmax at steady state for riociguat and its metabolite M-1 (BAY60-4552)
Aeur(0-7) | Pre-dose and up to 7 hours post-dose
  Amount of drug excreted via urine from zero to 7 hours after administration for riociguat and its metabolite M-1 (BAY60-4552)
%Aeur(0-7) | Pre-dose and up to 7 hours post-dose
  Aeur(0-7) expressed as percent of dose administered for riociguat and its metabolite M-1 (BAY60-4552)
Urinary excretion (over 24 hours) of N-terminal cross-linking telopeptides of type I collagen (NTX) | From -01 to 16 Days
  Marker of bone resorption
Serum CTX | From -01 to 16 Days
  Marker of bone resorption
Serum N-terminal propeptide of type I collagen (PINP) | From -01 to 16 Days
  Marker of bone formation
Serum bone-specific alkaline phosphatase (bAP) | From -01 to 16 Days
  Marker of bone formation
Serum albumin, protein | From -01 to 16 Days
  Determination of albumin, protein in serum
Cyclic guanosine monophosphate (cGMP) | From -01 to 16 Days
  Determination of cGMP in plasma and urinary excretion (over 24 hours)
Calcium, sodium, potassium | From -01 to 16 Days
  Determination of calcium, sodium, potassium in serum and urinary excretion (over 24 hours)
Urine volume | From -01 to 16 Days
  Volume of urine excreted (over 24 hours)
Renin | From -01 to 16 Days
  Determination of plasma renin level
Creatinine clearance | From -01 to 16 Days
  For estimation of glomerular filtration rate
Serum osteocalcin | From -01 to 16 Days
  Determination of osteocalcin in serum
Creatinine | From -01 to 16 Days
  Determination of creatinine in serum and urinary excretion (over 24 hours)
Phosphate | From -01 to 16 Days
  Determination of phosphate in serum only
Parathyroid hormone (PTH) | From -01 to 16 Days
  Determination of PTH in serum only

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/